CLINICAL TRIAL: NCT06649292
Title: An Open, Randomized,Positive Control, Multicenter Phase III Clinical Study of SHR A1904 for Injection Compared With Investigator's Choice of Therapy in Claudin18.2 Positive Patients With Second-line Advanced or Metastatic Gastric or Gastroesophageal Junction Adenocarcinoma
Brief Title: SHR-A1904 Compared With Investigator's Choice of Therapy in Claudin18.2 Positive Patitens With Second-line Advanced or Metastatic Gastric or Gastroesophageal Junction Adenocarcinoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-A1904-302
Record Dates: First submitted 2024-10-17; First posted 2024-10-18 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-10

CONDITIONS: Second-line Advanced or Metastatic Gastric or Gastroesophageal Junction Adenocarcinoma
MeSH Terms: interventions — Paclitaxel; Docetaxel; Irinotecan

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group A: SHR-A1904 (Experimental)
  Interventions: Drug: SHR-A1904
- Treatment group B: Paclitaxel, Docetaxel, Irinotecan. (Active Comparator)
  Interventions: Drug: Paclitaxel, Docetaxel, Irinotecan

INTERVENTIONS:
Drug: SHR-A1904 — SHR-A1904
  Arms: Treatment group A: SHR-A1904
Drug: Paclitaxel, Docetaxel, Irinotecan — Paclitaxel, Docetaxel, Irinotecan
  Arms: Treatment group B: Paclitaxel, Docetaxel, Irinotecan.

SUMMARY:
The study evaluated the overall survival (OS) of SHR-A1904 versus investigator-selected treatment in second-line CLDN18.2-positive advanced GC/GEJC patients

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 75 years old (including boundary values)
2. Volunteer to participate in this clinical study and sign informed consent;
3. ECOG score 0-1;
4. Expected survival ≥3 months;
5. Gastric or Gastroesophageal Junction Adenocarcinoma;
6. positive CLDN18.2 expression in tumor tissue;
7. There is at least one measurable or evaluable lesion that meets the RECIST 1.1 criteria;
8. Adequate bone marrow and organ function.

Exclusion Criteria:

1. Received anti-tumor therapies such as chemotherapy, radiotherapy, biological therapy, targeted therapy, or immunotherapy within 4 weeks before the first dose of the study
2. HER2 posotive (IHC 3+ or IHC 2+/ISH +);
3. Toxicities caused by previous anticancer therapy were not recovered to CTCAE 5.0 Grade≤1;
4. Individuals with Leptomeningeal metastasis or Active brain metastases;
5. Individuals with a history of GI perforation or fistula, unstable GI bleeding;
6. Individuals with a history of severe cardiovascular and cerebrovascular diseases;
7. The researcher determined that there are other situations that are not suitable for participation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 524 (Estimated)
Dates: Start 2024-11-22 (Actual); Primary Completion 2027-09-20 (Estimated); Study Completion 2028-03-20 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | Until death, assessed up to approximately 2 years
  Measure description: Defined as time from randomization until the date of death due to any cause

SECONDARY OUTCOMES:
Progression-free survival (PFS) by investigator assessment | Until progression or death, assessed up to approximately 1 year
  Measure description: Defined as time from randomization until progression or death as assessed by the investigator
Objective response rate (ORR) by investigator assessment | Until progression, assessed up to approximately 1 year
  Measure description: Defined as percentage of participants who achieved a best overall response of complete response (CR) or partial response (PR) assessed by the investigator
Duration of response (DOR) by investigator assessment | Until progression or death, assessed up to approximately 1 year
  Measure description: Defined as the time from the first documented objective response (CR or PR) to the first documented disease progression or death assessed by the investigator
Disease control rate (DCR) by investigator assessment | Until progression, assessed up to approximately 1 year
  Measure description: Defined as percentage of participants who achieved a best overall response of complete response (CR), partial response (PR) or stable disease (SD) assessed by the investigator
Incidence and severity of adverse events (AEs)/serious adverse events (SAEs) | until to 90 days after the last dose，assessed up to approximately 2 years
  Measure description: Incidence and severity of adverse events (AEs)/serious adverse events (SAEs) graded by Common Terminology Criteria for Adverse Events (CTCAE) v5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided